CLINICAL TRIAL: NCT02578901
Title: American Trial Using Tranexamic Acid in Thrombocytopenia (A-TREAT)
Brief Title: American Trial Using Tranexamic Acid in Thrombocytopenia
Acronym: A-TREAT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Susanne May, Professor, Biostatistics, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: STUDY00003329; 1U01HL122272-01A1 (NIH)
Record Dates: First submitted 2015-10-15; First posted 2015-10-19 (Estimated); Results first posted 2021-03-24 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-02

CONDITIONS: Thrombocytopenia
Keywords: Thrombocytopenia; Tranexamic Acid; TXA; Chemotherapy induced thrombocytopenia
MeSH Terms: conditions — Thrombocytopenia | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tranexamic Acid (TXA) (Active Comparator): IV or PO administered after meeting inclusion/exclusion criteria
  Interventions: Drug: Tranexamic Acid
- Placebo (Placebo Comparator): IV Normal Saline or PO placebo pills administered after meeting inclusion/exclusion criteria
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tranexamic Acid — Doses will be given intravenous (IV) or orally (PO) per the discretion of the treating investigator. Doses are administered every 8 hours. When given IV, TXA 1.0 gram will be administered. When given PO, TXA 1.3 grams will be administered
  Other Names: TXA
  Arms: Tranexamic Acid (TXA)
Drug: Placebo — Doses will be given intravenous (IV) or orally (PO) per the discretion of the treating investigator. Doses are administered every 8 hours. When given IV, Normal Saline will be administered. When given PO, placebo pills will be administered
  Other Names: NS
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the usefulness of antifibrinolytic therapy with tranexamic acid (TXA) in preventing bleeding in patients who are thrombocytopenic due to primary bone marrow disorders or chemotherapy, immunotherapy and/or radiation therapy.

DETAILED DESCRIPTION:
The purpose of this study is to conduct a prospective, randomized, blinded, placebo controlled trial to evaluate the usefulness of antifibrinolytic therapy with tranexamic acid in preventing bleeding in patients who are thrombocytopenic due to primary bone marrow disorders or chemotherapy, immunotherapy and/or radiation therapy. The results of this study will change practice by providing evidence as to whether or not TXA is effective and safe treatment when used as an adjunct to platelet transfusion therapy in the thrombocytopenic patient.

ELIGIBILITY:
Inclusion criteria (all must be met):

* Must be ≥ 18 years of age
* Confirmed diagnosis of a hematologic malignancy or aplasia
* Undergoing or planned chemotherapy, immunotherapy, or hematopoietic stem cell transplantation
* Anticipated to have hypoproliferative thrombocytopenia resulting in a platelet count of ≤ 10,000/microliters for ≥ 5 days
* Able to provide informed consent and comply with treatment and monitoring, or having a Legally Authorized Representative (LAR)

Exclusion criteria (none can be present):

* Diagnosis of acute promyelocytic leukemia undergoing induction chemotherapy
* History of ITP, TTP or HUS
* Subjects receiving L-asparaginase as part of their current cycle of treatment
* Subjects with a past history or current diagnosis of arterial or venous thromboembolic disease including acute coronary syndrome, peripheral vascular disease and retinal arterial or venous thrombosis (except when a prior history of central line thrombosis has resolved)
* Subjects with a diagnosis/previous history of sinusoidal obstruction syndrome (also called veno-occlusive disease)
* Subjects receiving any pro-coagulant agents (e.g. DDAVP, recombinant Factor VIIa or Prothrombin Complex Concentrates (PCC) and/or an antifibrinolytic agent within 48 hours of enrollment, or with known hypercoagulable state
* Known inherited or acquired bleeding disorder including, but not limited to:

  * Acquired storage pool deficiency
  * Paraproteinemia with platelet inhibition
* Known inherited or acquired prothrombotic disorders, including antiphospholipid syndrome. Those with lupus anticoagulant or positive antiphospholipid serology without thrombosis are not excluded.
* Subjects receiving anticoagulant therapy or anti-platelet therapy (except when receiving prophylactic anticoagulant or low dose aspirin therapy for prophylaxis only with a plan to discontinue when the platelet count falls below 50,000)
* Patients with DIC according to the patient's physician
* Subjects with WHO Grade 2 bleeding or greater within 48 hours prior to activation
* Subjects requiring a platelet transfusion threshold > 10,000/microliters at time of randomization
* Subjects with anuria (defined as urine output < 10mls/hr over 24 hours)
* Subjects on dialysis
* Subjects with creatinine ≥5.7mg/dL
* Subjects who are pregnant or nursing or unwilling to use contraception during and for 30 days after taking the study drug (both males and females)
* Subjects enrolled in other trials involving platelet transfusions, anti-fibrinolytics, platelet growth factors or other pro-coagulant agents.
* Known allergy to tranexamic acid
* Having been previously randomized in this study at any stage of their treatment
* Subjects who are unwilling to accept blood or blood component transfusions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2020-03 (Actual); Study Completion 2020-06-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terry Gernsheimer, MD, Principal Investigator — University of Washington
Locations (3):
- United States (3):
  - University of North Carolina, Chapel Hill, North Carolina
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Anonymized public data set will be available after publication of primary results
Time Frame: Public use data will be available within 3 years after primary outcome completion. These will be available through NHLBI and the duration of their availability will be according to NHLBI biolincc protocols.
Access Criteria: The access criteria will be according to NHLBI biolincc protocols at the time of the request.
URL: https://biolincc.nhlbi.nih.gov/home/

REFERENCES:
- [Derived] Poston JN, Brown SP, Ilich A, Ginsburg AS, Herren H, El Kassar N, Jensen CE, Triulzi DJ, Key NS, May S, Gernsheimer TB. Fewer severe infections with tranexamic acid in patients with hematologic malignancies. Res Pract Thromb Haemost. 2024 Mar 1;8(2):102358. doi: 10.1016/j.rpth.2024.102358. eCollection 2024 Feb. PMID 38666065
- [Derived] Ilich A, Gernsheimer TB, Triulzi DJ, Herren H, Brown SP, Holle LA, Lucas AT, de Laat B, El Kassar N, Wolberg AS, May S, Key NS. Absence of hyperfibrinolysis may explain lack of efficacy of tranexamic acid in hypoproliferative thrombocytopenia. Blood Adv. 2023 Mar 28;7(6):900-908. doi: 10.1182/bloodadvances.2022008255. PMID 36044391

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tranexamic Acid (TXA) | Placebo
Started | 165 | 165
Completed | 145 | 144
Not Completed | 20 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tranexamic Acid (TXA) | Placebo | Total
Number analyzed (Participants) | 165 | 165 | 330
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.1 (13.0) | 54.3 (13.2) | 54.2 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 65 | 138
  Male | 92 | 100 | 192
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 4 | 6
  Asian | 3 | 9 | 12
  Native Hawaiian or Other Pacific Islander | 2 | 3 | 5
  Black or African American | 11 | 12 | 23
  White | 141 | 129 | 270
  More than one race | 1 | 5 | 6
  Unknown or Not Reported | 5 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Bleeding Within 30 Days
Description: Proportion of patients with bleeding of WHO grade 2 or above, over the study period of 30 days after activation of study drug.
Time Frame: 30 days after activation of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Tranexamic Acid (TXA) | Placebo
Number analyzed (Participants) | 145 | 144
Participants | 73 | 78

2. Secondary Outcome: Number of Platelet Transfusions
Description: Number of platelet transfusions per patient during the first 30 days post prescription activation of study drug
Time Frame: 30 days after activation of study drug
Measure: Mean (Standard Deviation); unit: platelet transfusions
Arm/Group | Tranexamic Acid (TXA) | Placebo
Number analyzed (Participants) | 165 | 165
platelet transfusions | 7.7 (8.7) | 7.6 (10.1)

3. Secondary Outcome: Number of Days Alive and Without WHO Grade 2 Bleeding
Description: Number of days alive and without WHO grade 2 bleeding or greater during the first 30 days post activation of study drug
Time Frame: during the first 30 days post activation of study drug
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Tranexamic Acid (TXA) | Placebo
Number analyzed (Participants) | 136 | 132
days | 28.1 (3.7) | 27.7 (4.7)

ADVERSE EVENTS:
Time Frame: 120 days after activation
Arm/Group | Tranexamic Acid (TXA) | Placebo
All-Cause Mortality (participants affected / at risk) | 19/163 | 19/163
Serious Adverse Events (participants affected / at risk) | 123/163 | 110/163
Other Adverse Events (participants affected / at risk) | 161/163 | 161/163
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tranexamic Acid (TXA) (N=163) | Placebo (N=163)
Febrile neutropenia (Blood and lymphatic system disorders) | 40 | 36
Other blood/lymph disorder (Blood and lymphatic system disorders) | 2 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 1
Spleen disorder (Blood and lymphatic system disorders) | 0 | 1
Hemolysis (Blood and lymphatic system disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 10 | 9
Other cardiac (Cardiac disorders) | 3 | 4
Atrial fibrillation (Cardiac disorders) | 2 | 3
Atrial flutter (Cardiac disorders) | 2 | 1
Cardiac arrest (Cardiac disorders) | 1 | 1
Ventricular arrhythmia (Cardiac disorders) | 1 | 1
Pericardial effusion (Cardiac disorders) | 0 | 2
Heart failure (Cardiac disorders) | 1 | 1
Palpitations (Cardiac disorders) | 0 | 2
Myocardial infarction (Cardiac disorders) | 0 | 1
RV dysfunction (Cardiac disorders) | 1 | 0
Chest pain - cardiac (Cardiac disorders) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 0
Mitral valve disease (Cardiac disorders) | 1 | 0
Tricuspid valve disease (Cardiac disorders) | 1 | 0
Other congenital (Congenital, familial and genetic disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 3
Ear pain (Ear and labyrinth disorders) | 2 | 0
Other (Ear and labyrinth disorders) | 0 | 1
Blurred vision (Eye disorders) | 1 | 3
Other eye disorder (Eye disorders) | 2 | 2
Eye pain (Eye disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 27 | 16
Diarrhea (Gastrointestinal disorders) | 8 | 11
Abdominal pain (Gastrointestinal disorders) | 8 | 11
Vomiting (Gastrointestinal disorders) | 9 | 7
Constipation (Gastrointestinal disorders) | 10 | 4
Other gastrointestinal (Gastrointestinal disorders) | 4 | 6
Mucositis oral (Gastrointestinal disorders) | 4 | 3
Dyspepsia (Gastrointestinal disorders) | 2 | 5
Dysphagia (Gastrointestinal disorders) | 2 | 3
Esophageal pain (Gastrointestinal disorders) | 2 | 3
Rectal pain (Gastrointestinal disorders) | 4 | 0
Dry mouth (Gastrointestinal disorders) | 3 | 1
Ascites (Gastrointestinal disorders) | 1 | 2
Bloating (Gastrointestinal disorders) | 1 | 1
Hemorrhoids (Gastrointestinal disorders) | 2 | 0
Rectal ulcer (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Typhlitis (Gastrointestinal disorders) | 1 | 0
Rectal fistula (Gastrointestinal disorders) | 0 | 1
Rectal hemorrhage (Gastrointestinal disorders) | 1 | 0
Gastroesoph reflux disease (Gastrointestinal disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Oral pain (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 17 | 15
Fever (General disorders) | 12 | 12
Edema limbs (General disorders) | 7 | 13
Infusion related reaction (General disorders) | 3 | 5
Other general disorder (General disorders) | 3 | 2
Pain (General disorders) | 1 | 3
Chills (General disorders) | 0 | 4
Non-cardiac chest pain (General disorders) | 0 | 4
Multi-organ failure (General disorders) | 0 | 2
Edema face (General disorders) | 1 | 1
Malaise (General disorders) | 1 | 0
Neck edema (General disorders) | 1 | 0
Facial pain (General disorders) | 1 | 0
Other hepatobiliary (Hepatobiliary disorders) | 2 | 2
Hepatic failure (Hepatobiliary disorders) | 0 | 2
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Other immune disorder (Immune system disorders) | 18 | 12
Allergic reaction (Immune system disorders) | 1 | 0
Other infection (Infections and infestations) | 19 | 22
Sepsis (Infections and infestations) | 5 | 10
Lung infection (Infections and infestations) | 2 | 8
Sinusitis (Infections and infestations) | 3 | 5
Upper respiratory infection (Infections and infestations) | 4 | 3
Urinary tract infection (Infections and infestations) | 4 | 1
Skin infection (Infections and infestations) | 2 | 3
Abdominal infection (Infections and infestations) | 0 | 1
Papulopustular rash (Infections and infestations) | 0 | 1
Meningitis (Infections and infestations) | 0 | 1
Catheter related infection (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 4 | 2
Other injury (Injury, poisoning and procedural complications) | 3 | 3
Bruising (Injury, poisoning and procedural complications) | 3 | 0
Gastric anastomotic leak (Injury, poisoning and procedural complications) | 0 | 1
ALT increased (Investigations) | 1 | 4
Creatinine increased (Investigations) | 3 | 2
Weight gain (Investigations) | 3 | 2
AST increased (Investigations) | 1 | 3
Blood bilirubin increased (Investigations) | 1 | 2
Other investigation abnormal (Investigations) | 1 | 2
Urine output decreased (Investigations) | 1 | 2
Weight loss (Investigations) | 0 | 2
Alk phos increased (Investigations) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 11 | 5
Other metabolism disorder (Metabolism and nutrition disorders) | 4 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 4 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 3 | 2
Acidosis (Metabolism and nutrition disorders) | 1 | 3
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Hypernatremia (Metabolism and nutrition disorders) | 0 | 2
Hypoglycemia (Metabolism and nutrition disorders) | 2 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 1
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 1
Iron overload (Metabolism and nutrition disorders) | 0 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 3
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Other musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Joint ROM decreased (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Other neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Headache (Nervous system disorders) | 16 | 10
Dizziness (Nervous system disorders) | 9 | 5
Other nervous sys disorder (Nervous system disorders) | 3 | 5
Paresthesia (Nervous system disorders) | 4 | 2
Syncope (Nervous system disorders) | 3 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 1
Intracranial hemorrhage (Nervous system disorders) | 1 | 2
Encephalopathy (Nervous system disorders) | 0 | 3
Seizure (Nervous system disorders) | 1 | 1
Ataxia (Nervous system disorders) | 1 | 1
Dysgeusia (Nervous system disorders) | 2 | 0
Tremor (Nervous system disorders) | 1 | 1
Akathisia (Nervous system disorders) | 0 | 1
Ischemia cerebrovascular (Nervous system disorders) | 1 | 0
Transient ischemic attacks (Nervous system disorders) | 1 | 0
Stroke (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Dysphasia (Nervous system disorders) | 0 | 1
Dysesthesia (Nervous system disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 0 | 1
Vasovagal reaction (Nervous system disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 11 | 7
Other psychiatric disorder (Psychiatric disorders) | 4 | 2
Anxiety (Psychiatric disorders) | 2 | 3
Depression (Psychiatric disorders) | 3 | 1
Delirium (Psychiatric disorders) | 1 | 2
Confusion (Psychiatric disorders) | 0 | 3
Restlessness (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 7 | 6
Other renal disorder (Renal and urinary disorders) | 5 | 2
Urinary frequency (Renal and urinary disorders) | 2 | 2
Hematuria (Renal and urinary disorders) | 1 | 1
Renal calculi (Renal and urinary disorders) | 0 | 2
Urinary incontinence (Renal and urinary disorders) | 0 | 2
Urinary retention (Renal and urinary disorders) | 1 | 0
Urinary urgency (Renal and urinary disorders) | 0 | 1
Other reproductive sys disorder (Reproductive system and breast disorders) | 3 | 3
Testicular pain (Reproductive system and breast disorders) | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10 | 10
Other respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 8 | 11
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 10 | 7
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 7
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 | 7
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Apnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 | 12
Other skin disorder (Skin and subcutaneous tissue disorders) | 5 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 4
Dry skin (Skin and subcutaneous tissue disorders) | 4 | 3
Skin ulceration (Skin and subcutaneous tissue disorders) | 4 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 3
Purpura (Skin and subcutaneous tissue disorders) | 1 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 2
Skin induration (Skin and subcutaneous tissue disorders) | 0 | 1
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1
Hypotension (Vascular disorders) | 13 | 11
Hypertension (Vascular disorders) | 6 | 7
Thromboembolic event (Vascular disorders) | 3 | 4
Flushing (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tranexamic Acid (TXA) (N=163) | Placebo (N=163)
Febrile neutropenia (Blood and lymphatic system disorders) | 81 | 75
Sinus tachycardia (Cardiac disorders) | 70 | 65
Sinus bradycardia (Cardiac disorders) | 14 | 8
Other cardiac (Cardiac disorders) | 10 | 6
Other (Ear and labyrinth disorders) | 9 | 4
Blurred vision (Eye disorders) | 18 | 12
Other eye disorder (Eye disorders) | 9 | 18
Fatigue (General disorders) | 100 | 102
Edema limbs (General disorders) | 65 | 64
Chills (General disorders) | 28 | 27
Infusion related reaction (General disorders) | 26 | 29
Fever (General disorders) | 25 | 28
Other general disorder (General disorders) | 26 | 24
Pain (General disorders) | 23 | 15
Injection site reaction (General disorders) | 15 | 17
Non-cardiac chest pain (General disorders) | 16 | 9
Localized edema (General disorders) | 11 | 12
Edema face (General disorders) | 11 | 11
Diarrhea (Gastrointestinal disorders) | 114 | 112
Nausea (Gastrointestinal disorders) | 95 | 91
Abdominal pain (Gastrointestinal disorders) | 68 | 55
Mucositis oral (Gastrointestinal disorders) | 58 | 63
Vomiting (Gastrointestinal disorders) | 65 | 56
Constipation (Gastrointestinal disorders) | 43 | 52
Other gastrointestinal (Gastrointestinal disorders) | 36 | 42
Dry mouth (Gastrointestinal disorders) | 20 | 25
Dyspepsia (Gastrointestinal disorders) | 26 | 17
Oral pain (Gastrointestinal disorders) | 15 | 15
Gastroesoph reflux disease (Gastrointestinal disorders) | 13 | 14
Bloating (Gastrointestinal disorders) | 14 | 11
Rectal pain (Gastrointestinal disorders) | 12 | 12
Hemorrhoids (Gastrointestinal disorders) | 16 | 7
Fecal incontinence (Gastrointestinal disorders) | 6 | 11
Abdominal distension (Gastrointestinal disorders) | 9 | 7
Other hepatobiliary (Hepatobiliary disorders) | 11 | 8
Other immune disorder (Immune system disorders) | 21 | 14
Other infection (Infections and infestations) | 52 | 52
Skin infection (Infections and infestations) | 14 | 22
Sinusitis (Infections and infestations) | 13 | 15
Lung infection (Infections and infestations) | 14 | 6
Other injury (Injury, poisoning and procedural complications) | 9 | 13
ALT increased (Investigations) | 27 | 19
AST increased (Investigations) | 22 | 16
Weight gain (Investigations) | 10 | 12
Blood bilirubin increased (Investigations) | 15 | 7
Anorexia (Metabolism and nutrition disorders) | 69 | 65
Hyperglycemia (Metabolism and nutrition disorders) | 30 | 23
Other metabolism disorder (Metabolism and nutrition disorders) | 25 | 22
Hypokalemia (Metabolism and nutrition disorders) | 24 | 19
Hypomagnesemia (Metabolism and nutrition disorders) | 15 | 18
Hyponatremia (Metabolism and nutrition disorders) | 13 | 11
Hypophosphatemia (Metabolism and nutrition disorders) | 9 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 42 | 44
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 32 | 35
Back pain (Musculoskeletal and connective tissue disorders) | 36 | 28
Pain in extremity (Musculoskeletal and connective tissue disorders) | 32 | 30
Neck pain (Musculoskeletal and connective tissue disorders) | 12 | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 11
Bone pain (Musculoskeletal and connective tissue disorders) | 8 | 9
Other musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 4 | 10
Headache (Nervous system disorders) | 66 | 67
Dizziness (Nervous system disorders) | 38 | 38
Dysgeusia (Nervous system disorders) | 34 | 30
Tremor (Nervous system disorders) | 16 | 19
Peripheral sensory neuropathy (Nervous system disorders) | 14 | 14
Paresthesia (Nervous system disorders) | 9 | 15
Insomnia (Psychiatric disorders) | 37 | 49
Anxiety (Psychiatric disorders) | 30 | 33
Confusion (Psychiatric disorders) | 13 | 11
Depression (Psychiatric disorders) | 10 | 11
Other psychiatric disorder (Psychiatric disorders) | 9 | 8
Other renal disorder (Renal and urinary disorders) | 27 | 26
Urinary frequency (Renal and urinary disorders) | 19 | 13
Acute kidney injury (Renal and urinary disorders) | 8 | 17
Urinary urgency (Renal and urinary disorders) | 10 | 11
Urinary incontinence (Renal and urinary disorders) | 9 | 8
Urinary retention (Renal and urinary disorders) | 9 | 5
Other reproductive sys disorder (Reproductive system and breast disorders) | 9 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 38 | 53
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 40 | 41
Other respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 33 | 33
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 32 | 33
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 24 | 31
Productive cough (Respiratory, thoracic and mediastinal disorders) | 26 | 21
Sore throat (Respiratory, thoracic and mediastinal disorders) | 20 | 20
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 23 | 17
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 17 | 16
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 15 | 16
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 | 18
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 12 | 11
Wheezing (Respiratory, thoracic and mediastinal disorders) | 14 | 9
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 9 | 8
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 71 | 62
Other skin disorder (Skin and subcutaneous tissue disorders) | 40 | 53
Pruritus (Skin and subcutaneous tissue disorders) | 41 | 48
Dry skin (Skin and subcutaneous tissue disorders) | 20 | 31
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 13 | 16
Skin ulceration (Skin and subcutaneous tissue disorders) | 17 | 10
Hypotension (Vascular disorders) | 53 | 56
Hypertension (Vascular disorders) | 50 | 56

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2018-05-07): https://cdn.clinicaltrials.gov/large-docs/01/NCT02578901/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-03): https://cdn.clinicaltrials.gov/large-docs/01/NCT02578901/SAP_001.pdf
  • Informed Consent Form (2016-06-24): https://cdn.clinicaltrials.gov/large-docs/01/NCT02578901/ICF_002.pdf